CLINICAL TRIAL: NCT02343913
Title: Simplifying Menstrual Regulation (MR): Exploring the Role of At-home Semi-quantitative Pregnancy Tests for Follow-up to Menstrual Regulation Service Provision in Pakistan: Post Abortion Care (PAC)
Brief Title: Simplifying Menstrual Regulation (MR): Post Abortion Care in Pakistan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gynuity Health Projects (Other)
Collaborators: Family Planning Association Pakistan (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 6005a
Record Dates: First submitted 2015-01-16; First posted 2015-01-22 (Estimated); Last update posted 2015-03-03 (Estimated); Status verified 2015-03

CONDITIONS: Medical Abortion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PAC checklist (Experimental): Pictorial checklist which illustrates these signs and symptoms
  Interventions: Device: PAC checklist

INTERVENTIONS:
Device: PAC checklist

SUMMARY:
This study is an additional component of protocol 6005, titled Simplifying Menstrual Regulation (MR): Exploring the role of at-home semi-quantitative pregnancy tests for follow-up to menstrual regulation service provision in Pakistan. The study seeks to pilot a self-assessment checklist that will help women, who receive medical services for incomplete abortion, correctly identify warning signs and symptoms and determine whether to return to the clinic. The checklist can serve as a useful resource to help with the timely identification of women who need additional care and can help streamline service delivery. In addition, this study will provide important data on the role of misoprostol at varying levels of health services offering an array of treatments for incomplete abortion.

ELIGIBILITY:
Inclusion Criteria:

* Vaginal bleeding during pregnancy
* Open cervical os.
* No signs of severe infection, defined as at least one of the following of: 1) foul smelling discharge, 2) fever > 38 degrees C , 3) uterine tenderness
* No hemodynamic disturbances (pulse >110/min and systolic bp <100)

Exclusion Criteria:

* Suspected to have an ectopic pregnancy
* Unable to provide informed consent

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 329 (Actual)
Dates: Start 2014-06; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Identify symptoms | 1 week
  Proportion of women able to use a checklist to correctly identify any signs and symptoms that warrant immediate return to the clinic and additional care

SECONDARY OUTCOMES:
Acceptability of treatment | 1 week
  Proportion of women who find the treatment of 400 sublingual misoprostol for incomplete abortion acceptable and satisfactory.
Uptake of contraceptive use | 1 week
  Proportion of women who receive a contraceptive method after receipt of 400 sublingual misoprostol

CONTACTS AND LOCATIONS:
Overall Officials: Dina Abbas, MPH, Principal Investigator — Gynuity Health Projects; Anjum Rizvi, MBBS, MHA, Principal Investigator — Rahnuma FPAP; Asifa Khanum, MPhil, MSc, Principal Investigator — Rahnuma FPAP; Beverly Winikoff, MD, MPH, Principal Investigator — Gynuity Health Projects
Locations (15):
- Pakistan (15):
  - Bhagwal Service Delivery Clinic, Bhagwal, Chakwal
  - Chakumra Service Delivery Clinic, Chakumra, Chakwal
  - Karrila Service Delivery Clinic, Karrila, Chakwal
  - Khanpur Service Delivery Clinic, Khanpur, Chakwal
  - Chak 128 GB Service Delivery Clinic, Faisalabad, Faisalabad
  - BagaSher Service Delivery Clinic, BagaSher, Muzaffargarh
  - Dasrat Colony Service Delivery Clinic, Dasrat Colony, Muzaffargarh
  - Fazal Nagal Service Delivery Clinic, Fazal Nagal, Muzaffargarh
  - Bahari Colony Service Delivery Clinic, Bahari Colony, Rawalpindi
  - DhokeHasso Service Delivery Clinic, DhokeHasso, Rawalpindi
  - Model Clinic Chakwal, Chakwal
  - Model Clinic Faisalabad, Faisalabad
  - Family Health Hospital, Islamabad
  - Family Health Hospital, Lahore
  - Sabe wala clinic, Muzaffargarh